CLINICAL TRIAL: NCT00107744
Title: Clinical Trial of Protein and Blood Pressure
Acronym: ProBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H0330; R01HL068057 (NIH)
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2018-06

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: Blood Pressure; Lipids; Dietary Protein
MeSH Terms: conditions — Hypertension; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: The trial participants were assigned to take 40 g/d soy protein, milk protein, or carbohydrate supplementation each for 8 weeks in a random order. A 3-week washout period was implemented between the interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization assignment list was generated by a computer program that could only be accessed by the study data coordinator. Apart from the data coordinator, all research personnel, including investigators, study coordinators, and BP technicians, and the study participants were unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Soy protein-milk protein-carbohydrate (Active Comparator): Participants received 40 grams of soy protein daily for 8 weeks, 40 grams of milk protein daily for 8 weeks, and 40 grams of carbohydrate daily for 8 weeks.
  Interventions: Dietary Supplement: Soy protein-milk protein-carbohydrate
- Milk protein-carbohydrate-soy protein (Active Comparator): Participants received 40 grams of milk protein daily for 8 weeks, 40 grams of carbohydrate daily for 8 weeks, and 40 grams of soy protein daily for 8 weeks.
  Interventions: Dietary Supplement: Milk protein-carbohydrate-soy protein
- Carbohydrate-soy protein-milk protein (Active Comparator): Participants received 40 grams of complex carbohydrate daily for 8 weeks, 40 grams of soy protein daily for 8 weeks, and 40 grams of milk protein daily for 8 weeks.
  Interventions: Dietary Supplement: Carbohydrate-soy protein-milk protein

INTERVENTIONS:
Dietary Supplement: Soy protein-milk protein-carbohydrate — 40 grams of soy protein per day for 8 weeks, 40 grams of milk protein per day for 8 weeks, and 40 grams of carbohydrate per day for 8 weeks
  Arms: Soy protein-milk protein-carbohydrate
Dietary Supplement: Milk protein-carbohydrate-soy protein — 40 grams of milk protein per day for 8 weeks, 40 grams of carbohydrate per day for 8 weeks, 40 grams of soy protein per day for 8 weeks.
  Arms: Milk protein-carbohydrate-soy protein
Dietary Supplement: Carbohydrate-soy protein-milk protein — 40 grams of carbohydrate per day for 8 weeks, 40 grams of soy protein per day for 8 weeks, 40 grams of milk protein per day for 8 weeks.
  Arms: Carbohydrate-soy protein-milk protein

SUMMARY:
The purpose of this randomized, double-blind, controlled trial is to examine the effect of soybean protein supplementation on blood pressure in persons with prehypertension or stage-1 hypertension.

DETAILED DESCRIPTION:
Background: Epidemiologic studies suggest that vegetable protein intake is inversely related to blood pressure.

Objectives: To examine the effect of soybean protein supplementation on blood pressure in persons with prehypertension or stage-1 hypertension

Design: Randomized, double-blind, controlled trial

Study Participants: 350 participants, aged 35-64 years, with an initial untreated systolic blood pressure of 130-159 mmHg and/or diastolic blood pressure of 80-99 mmHg

Intervention: Study participants will be randomly assigned to take 40-grams of isolated soybean protein supplements per day or complex carbohydrate control for 12 weeks.

Outcomes: Blood pressure measurements will be obtained using random-zero sphygmomanometers at baseline and during the trial at weeks 6 and 12. Net changes in systolic and diastolic blood pressure before and after the intervention is the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic BP of 120 to 159 mm Hg and diastolic BP of 80 to 95 mm Hg (average of 6 measurements at 2 screening visits)
2. Willing to participate in all aspects of the study

Exclusion Criteria:

1. Consumption of dietary protein greater than or equal to 1.63 grams/kg per day, as determined by two 24-hour dietary recalls
2. Stage-2 or higher severe hypertension (systolic BP greater than or equal to 160 mm Hg and/or diastolic BP greater than or equal to 95 mm Hg)
3. Use of antihypertensive medications or medications that affect BP
4. History of clinical heart disease (e.g., angina/heart attack, coronary revascularization, heart failure, stroke/transient ischemic attack, peripheral arterial disease)
5. Kidney disease (serum creatinine level greater than or equal to 1.7 mg/dL for men and greater than or equal to 1.5 mg/dL for women)
6. Current hypercholesterolemia (fasting serum total cholesterol greater than or equal to 240 mg/dL) or use of cholesterol-lowering medications
7. Current diabetes (fasting serum glucose greater than or equal to 126 mg/dL) or use of insulin or oral hypoglycemic agents
8. Severe obesity (body mass index greater than or equal to 40 kg/m²)
9. Current use of prescription weight loss medications, underwent weight loss surgery, and/or experienced weight loss greater than 15 pounds within the 6 months prior to study entry
10. Cancer (except non-melanoma skin cancer) that required treatment during the year prior to study entry
11. Consumption of more than 14 alcoholic beverages per week
12. Current participation in another medical study
13. Consumption of milk or soy protein greater than or equal to the 90th percentile of intake in the U.S. general population
14. Has another member of the household participating in the study
15. Study employees or living with study employees
16. Allergy or intolerance to soy protein or milk protein products
17. Allergy to aspartame
18. Plans to move out of the study area (greater than or equal to 50 miles from the study site) and has difficulty coming to the study site
19. Inability or unwillingness to cooperate during the screening visits
20. Poor compliance during the screening period (intake of less than 85% of supplements)
21. Pregnant or plans to become pregnant during the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Study Chair — Tulane University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Result] He J, Wofford MR, Reynolds K, Chen J, Chen CS, Myers L, Minor DL, Elmer PJ, Jones DW, Whelton PK. Effect of dietary protein supplementation on blood pressure: a randomized, controlled trial. Circulation. 2011 Aug 2;124(5):589-95. doi: 10.1161/CIRCULATIONAHA.110.009159. Epub 2011 Jul 18. PMID 21768541
- [Result] Wofford MR, Rebholz CM, Reynolds K, Chen J, Chen CS, Myers L, Xu J, Jones DW, Whelton PK, He J. Effect of soy and milk protein supplementation on serum lipid levels: a randomized controlled trial. Eur J Clin Nutr. 2012 Apr;66(4):419-25. doi: 10.1038/ejcn.2011.168. Epub 2011 Sep 28. PMID 21952693
- [Result] Rebholz CM, Reynolds K, Wofford MR, Chen J, Kelly TN, Mei H, Whelton PK, He J. Effect of soybean protein on novel cardiovascular disease risk factors: a randomized controlled trial. Eur J Clin Nutr. 2013 Jan;67(1):58-63. doi: 10.1038/ejcn.2012.186. Epub 2012 Nov 28. PMID 23187956
- [Derived] Sun Y, Zhang R, Tian L, Liu T, Pan Y, Sun X, Huang Z, Fan J, Chen J, Zhang K, Li S, Chen W, Bazzano LA, He J, Bundy JD, Kelly TN, Li C. Associations of plasma inosine with lipid parameters in a biracial community cohort. Clin Nutr. 2025 Dec;55:113-123. doi: 10.1016/j.clnu.2025.10.011. Epub 2025 Oct 29. PMID 41202661

RESULTS

PARTICIPANT FLOW:
Period: Intervention 1 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate | Milk Protein-carbohydrate-soy Protein | Carbohydrate-soy Protein-milk Protein
Started | 117 | 117 | 118
Completed | 101 | 104 | 101
Not Completed | 16 | 13 | 17
Period: Intervention 2 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate | Milk Protein-carbohydrate-soy Protein | Carbohydrate-soy Protein-milk Protein
Started | 101 | 104 | 101
Completed | 93 | 92 | 88
Not Completed | 8 | 12 | 13
Period: Intervention 3 (8 Weeks)
Arm/Group | Soy Protein-milk Protein-carbohydrate | Milk Protein-carbohydrate-soy Protein | Carbohydrate-soy Protein-milk Protein
Started | 93 | 92 | 88
Completed | 93 | 92 | 88
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized to this three-phase cross-over trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Soy Protein-milk Protein-carbohydrate | Milk Protein-carbohydrate-soy Protein | Carbohydrate-soy Protein-milk Protein | Total
Number analyzed (Participants) | 117 | 117 | 118 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.5) | 46.7 (10.7) | 48.1 (8.7) | 47.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 50 | 147
  Male | 69 | 68 | 68 | 205
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 39 | 38 | 44 | 121
  White | 78 | 79 | 74 | 231
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 117 | 118 | 352
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 127.2 (9.3) | 126.7 (11.0) | 126.1 (9.7) | 126.7 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Systolic Blood Pressure at 8 Weeks
Description: The change of systolic blood pressure was calculated as the mean of 6 blood pressure values from two 8-week visits minus the mean of 6 values from 2 baseline visits within each intervention phase. At each visit, 3 BP values were measured with a Hawksley random-zero sphygmomanometer by trained and certified observers who were masked to group assignment. BP readings were taken from the right arm with appropriately sized cuffs after the participant had been seated quietly for 5 minutes. The participant was instructed not to eat, smoke, drink alcohol, or exercise for at least 30 minutes before their BP measurements.
Time Frame: Baseline and 8 Weeks
Population: We conducted analysis according to intention-to-treat principle. All participants with data were included in analysis.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Soy Protein Supplementation: Cross-over analysis of soy protein supplementation
- Milk Protein Supplementation; Carbohydrate Supplementation: Cross-over analysis of milk protein supplementation
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 284 | 286 | 287
mmHg | -1.5 [-2.4 to -0.6] | -1.8 [-2.7 to -1.0] | 0.5 [-0.4 to 1.3]

2. Secondary Outcome: Change From Baseline in Serum LDL-cholesterol at 8 Weeks
Description: Change in serum LDL-cholesterol was calculated as LDL-cholesterol at 8 weeks minus LDL-cholesterol at baseline. Over-night fasting serum LDL-cholesterol was measured with an enzymatic method.
Time Frame: Baseline and 8 Weeks
Population: All participants with lipid data
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 284 | 286 | 287
mg/dL | -3.97 [-7.63 to -0.31] | -2.56 [-5.40 to 0.28] | -1.41 [-4.24 to 1.42]

3. Secondary Outcome: Body Weight at 8 Weeks
Description: Body weight was measured by trained staff using a standard protocol at week 8.
Time Frame: Baseline and 8 Weeks
Population: All participants with body weight measures at each intervention phase
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
Number analyzed (Participants) | 284 | 286 | 287
kg | 86.2 [84.4 to 88.0] | 86.6 [84.9 to 88.4] | 86.7 [84.9 to 88.5]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 24 weeks
Description: This is a three-phase cross-over trial: 284 participants completed soy protein supplementation, 286 completed milk protein supplementation, and 287 completed carbohydrate supplementation.
Arm/Group | Soy Protein Supplementation | Milk Protein Supplementation | Carbohydrate Supplementation
All-Cause Mortality (participants affected / at risk) | 0/352 | 0/352 | 0/352
Serious Adverse Events (participants affected / at risk) | 0/352 | 0/352 | 0/352
Other Adverse Events (participants affected / at risk) | 0/352 | 0/352 | 0/352

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes